CLINICAL TRIAL: NCT06843733
Title: Feasibility Study of Mixed Reality Exergame on Performance and Cortical Outcomes in Healthy Older Adults and People with Mild Cognitive Impairment
Brief Title: Feasibility Study of Mixed Reality Exergame on Performance and Cortical Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Rommanee Rojasavastera, Principal Investigator, Faculty of Physical Therapy, Mahidol University, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MU-CIRB 2024/060.2102
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Executive Dysfunction; Mild Cognitive Impairment (MCI)
Keywords: Feasibility study; Mixed reality; Mild cognitive impairment; Executive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mild cognitive impairment (Experimental)
  Interventions: Other: Mixed reality exergame; Other: Education
- Healthy older adults (Other)
  Interventions: Other: Mixed reality exergame

INTERVENTIONS:
Other: Mixed reality exergame — The participants will play the Balloon Popping game using Hololens2 (Mixed reality glasses) for one hour. The objective of this game will be to pop all the virtual balloons, focusing on training different executive functions such as inhibitory control and cognitive flexibility. When a participant raises a finger in the air, a virtual needle will appear. After that, the participant will move their finger towards a balloon. Successful contact with a balloon will be indicated by the sound of a pop and the visual effect of confetti.
Other: Education — The participants will seat on a chair and watch video clip about MCI and dementia for one hour.
  Arms: Mild cognitive impairment

SUMMARY:
The executive dysfunctions are a problem in individuals with MCI which predict conversion to dementia and is positively related to physical activity level. Previous studies found that exercise can prevent executive and physical dysfunctions for people with MCI. However, the motivation is a critical factor in supporting a sustainable exercise. Exergame is combination of exercise and video game. Enjoyment during playing an exergame can support the exercise motivation. Therefore, we will explore the feasibility of using MR exergame in people with MCI.

ELIGIBILITY:
Inclusion Criteria

* Healthy group: 1) MoCA score > 24; 2) Independent walking without using gait aids; 3) No diagnosis of the dementia by clinician.
* MCI group: 1) MoCA score between 16 to 24; 2) Independent walking without using gait aids.

Exclusion Criteria:

* Uncontrolled high blood pressure (more than 140/90 mmHg)
* Hemodialysis
* Have clinical diagnosis of the disease or symptoms that could influence the performance assessments such as arthritis or severe hand pain which reports by participants and the testing by physiotherapist before testing.
* History of neurological disorder, such as stroke or other neurodegenerative disorder
* Taking medicine which affected to functional movement.
* Unable to follow study protocol.
* Uncorrected visual or hearing impairment.
* Positive screening for contraindication of TMS which will be confirmed by TMS screening questionnaire such as uncontrolled seizures.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual attention and task switching | before and immediately after intervention
  Trail Making Test
Inhibitory control | before and immediately after intervention
  Color-Word Stroop Test
Single-task performance | before and immediately after intervention
  Box and Block Test
Dual-task performance | before and immediately after intervention
  Box and Block with Serial Sevens Test
Cortical outcomes | before and immediately after intervention
  Transcranial magnetic stimulation was used for measuring the cortical outcomes, which consist of resting motor threshold, input-output curve of motor evoked potentials recruitment and cortical silent period.
Usability | immediately after Mixed reality exergaming
  System usability scale questionnaire was used for measuring the usability of mixed reality exergame. It consists of 10-item, which are typically rated on a five-point scale. A higher SUS score generally indicates better usability.
Motivation | immediately after Mixed reality exergaming
  Intrinsic Motivation Inventory was used for measuring the motivation. It rated on seven-point scale. Higher IMI scores reflect higher levels of motivation.
Adverse side effects | immediately after Mixed reality exergaming
  Cybersickness in Virtual Reality Questionnaire was used for assessing cybersickness symptoms, including nausea, vestibular, and oculomotor. The total score is the sum of the three sub-scores. Each question is presented on a 7-item Likert Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
We will share IPD when we receive the consent from participants.